CLINICAL TRIAL: NCT03042312
Title: PSMA-directed endoRadiothErapy of Castration-reSISTant Prostate Cancer (RESIST-PC). A Phase II Clinical Trial
Brief Title: Lutetium-177 (Lu177) Prostate-Specific Antigen (PSMA)-Directed EndoRadiotherapy
Acronym: RESIST-PC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was stopped before the target sample size was achieved.
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSMA-617-02; 133661 (Other: Original sponsor)
Record Dates: First submitted 2017-01-18; First posted 2017-02-03 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 177Lu-PSMA-617 (6.0 GBq) (Experimental): Repeated i.v. application of 6.0 GBq (gigabequerel)(+/- 10%, arm 1) every 8+/- 1 weeks; RLT until reaching four cycles or threshold maximum dose to the kidneys of 23 Gy as determined by dosimetry
  Interventions: Drug: 177Lu-PSMA-617
- 177Lu-PSMA-617 (7.4 GBq) (Experimental): Repeated i.v. application of 7.4 GBq (gigabequerel)(+/- 10%, arm 2) of drug every 8+/- 1 weeks; RLT until reaching four cycles or threshold maximum dose to the kidneys of 23 Gy as determined by dosimetry
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Lutetium (177Lu) -DOTA (1,4,7,10-tetra-azacyclododecane-N,N',N'',N'''-tetraacetic acid )-PSMA has three components: PSMA is the targeting vector , DOTA (1, 4, 7, 10-tetraazacyclododecane-1, 4, 7, 10-tetraacetic acid) is a radiometal chelator and a linking group, and 177Lu is the beta emitter that upon internalization delivers radiation to the nucleus of tumor cells to cause DNA damage. The targeting vector utilizes glu-urea-lys sequence which is an inhibitor capable of binding to the domain of PSMA. These components have been previously used in human subjects and in medical research.
  Other Names: Lu177 RLT

SUMMARY:
This was an open-label, multicenter, prospective trial to assess safety and efficacy of 177Lu-PSMA-617 in patients with metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
Upon inclusion patients were randomized in a 1:1 ratio into two treatment doses. Radioligand therapy (RLT) were performed by repeated intravenous (i.v.) injection of 6.0 gigabecquerel (GBq) (+/- 10%) or 7.4 GBq (+/- 10%) 177Lu-PSMA-617 every 8+/- 1 weeks until reaching four cycles or threshold maximum dose to the kidneys of 23 Gray (Gy). All doses after labeling were presented in buffered solution for i.v. injection.

In the initial plan for the study design a total of 200 patients with histologically proven prostate cancer and metastatic castration-resistant prostate cancer (mCRPC) were to be enrolled, however due to early stopping of enrollment only 71 patients were enrolled at time of data base lock. Each patient underwent a screening visit within 14 days prior to receiving study drug. Treatment was continued until either of the following conditions applied:

* Prostate-specific antigen (PSA)/radiographic progression at >= 12 weeks
* Completion of four RLT cycles
* 23 Gy kidney dose would be exceeded by the next cycle as estimated by dosimetry
* Patient withdrawal (e.g. appearance of intolerable adverse events).

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer proven by histopathology
2. Unresectable metastases
3. Progressive disease, both docetaxel naive and docetaxel treated.
4. Castration resistant disease with confirmed testosterone level ≤50 ng/ml under prior androgen deprivation therapy (ADT)
5. Positive 68Ga-PSMA-11 PET/CT (positron emission computed tomography ) or diagnostic 177Lu-PSMA-617 scintigraphy
6. ECOG 0-2
7. Sufficient bone marrow capacity as defined by WBC (white blood cell ) ≥2.500/μl, PLT (platelet) count ≥100.000/μl, Hb≥9.9 g/dl and ANC≥1500 mm3 for the first cycle and WBC≥2.000/ μl,PLT count ≥75.000/μl, Hb≥8.9 g/dl and ANC≥1000 mm3 for the subsequent cycles
8. Signing of the Informed Consent Form
9. Patients enrolling in this trail should have received either Enzalutamide or Abiraterone

Exclusion Criteria:

1. Less than 6 weeks since last myelosuppressive therapy (including Docetaxel, Cabazitaxel, 223Ra, 153Sm) or other radionuclide therapy.
2. Glomerular Filtration Rate (GFR) <40 ml/min
3. Serum creatinine > 1.5 ULN
4. AST and ALT>5xULN
5. Urinary tract obstruction or marked hydronephrosis
6. Diffuse bone marrow involvement confirmed by super-scans

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gafita A, Calais J, Grogan TR, Hadaschik B, Wang H, Weber M, Sandhu S, Kratochwil C, Esfandiari R, Tauber R, Zeldin A, Rathke H, Armstrong WR, Robertson A, Thin P, D'Alessandria C, Rettig MB, Delpassand ES, Haberkorn U, Elashoff D, Herrmann K, Czernin J, Hofman MS, Fendler WP, Eiber M. Nomograms to predict outcomes after 177Lu-PSMA therapy in men with metastatic castration-resistant prostate cancer: an international, multicentre, retrospective study. Lancet Oncol. 2021 Aug;22(8):1115-1125. doi: 10.1016/S1470-2045(21)00274-6. Epub 2021 Jul 8. PMID 34246328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in the USA
Period: Overall Study
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Started (All randomized participants were included in Intent-to-treat (ITT) population) | 28 | 43
Safety Population (The subset of patients in the ITT population who received at least one dose of randomized therapy.) | 23 | 41
Completed | 18 | 31
Not Completed | 10 | 12
Not completed — Administrative Reason | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Any occurrence of conditions which prevented the patient's participation in the study. | 4 | 2
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq) | Total
Number analyzed (Participants) | 28 | 43 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.1 (8.39) | 69.1 (8.62) | 70.3 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 43 | 71
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 0 | 1 | 1
  White | 26 | 41 | 67
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were collected from first dosing up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent. The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: From first dosing (Day 0) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent, up to 24 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 23 | 41
Participants
  Treatment-Emergent Adverse Events (TEAEs) | 22 | 39
  Serious TEAEs | 4 | 8
  Drug-related TEAEs | 20 | 37
  Serious drug-related TEAEs | 1 | 4
  TEAEs leading to reduction of Lu-PSMA-617 | 0 | 2
  TEAEs leading to discontinuation of Lu-PSMA-617 | 0 | 1
  TEAEs leading to death | 2 | 1

2. Primary Outcome: Number of Participants Achieving PSA Response at Week 12
Description: PSA response was defined as the proportion of patients who had a >= 50% decrease in PSA from Baseline at Week 12.
Time Frame: Week 12
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 14 | 25
Participants
  PSA Response (< 50% decline) | 5 | 8
  PSA Response (>= 50% decline) | 6 | 6
  PSA Response (Increase from Baseline) | 3 | 11

3. Secondary Outcome: Percent Change in PSA From Baseline to Week 12
Description: Percent change in PSA from Baseline to Week 12 was reported for participants who had a baseline and a week 12 valid assessments.
Time Frame: Week 12
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change in PSA
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 14 | 25
Percent change in PSA | -22.54 (75.513) | 92.15 (301.932)

4. Secondary Outcome: Maximum Percent Change in PSA Response
Description: Maximal baseline to follow-up PSA decline, at any time during or after therapy was evaluated in both treatment groups.
Time Frame: Every 6 weeks during the treatment and every 3 (+/- 1) months after last treatment until reaching endpoint or 24 months after the first treatment
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: PSA percent change
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 23 | 40
PSA percent change | -3.63 (95.394) | 8.75 (132.954)

5. Secondary Outcome: PSA Progression and Death Events
Description: PSA progression was defined as:
  1. For patients with PSA decline: PSA progression was defined as the date that a >= 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir was documented and confirmed by a second consecutive value obtained 3 or more weeks later. Rises in PSA within the first 12 weeks were ignored (PCWG3 Guidance),
  2. For patients without PSA decline: PSA progression was defined as a >= 25% increase from the baseline value along with an increase in absolute value of 2 ng/mL or more after 12 weeks of treatment.
Time Frame: Date of randomization to the date of first documented PSA progression or death, whichever occurs first, reported between day of first patient randomized up to 24 months after the first treatment
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 28 | 43
Participants
  Deaths without PSA progression | 2 | 2
  Participants with PSA progression, but who did not die | 11 | 17

6. Secondary Outcome: RECIST 1.1 Overall Response by Follow-up Assessment Visit
Description: For each follow-up imaging assessment by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target, non-target, and new lesions assessed by CT or MRI: the number of participants with an overall response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD).
  The timing of follow-up imaging assessments varied depending on how many RLT cycles a participant received. Therefore, regardless of when the imaging assessments occurred, each participant's first follow-up imaging was combined as Follow-up 1, each participant's second follow-up imaging was combined as Follow-up 2, each participant's third follow-up imaging was combined as Follow-up 3, and each participant's fourth follow-up imaging was combined as Follow-up 4.
Time Frame: Before 3rd radioligand therapy (RLT) cycle, and then every 3 (+/- 1) months after last treatment dose until disease progression or 24 months after the first treatment dose.
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 28 | 43
Participants
  Follow-up 1: number analyzed (Participants) | 11 | 21
  Follow-up 1: Complete Response | 1 | 1
  Follow-up 1: Partial Response | 3 | 4
  Follow-up 1: Stable Disease | 1 | 7
  Follow-up 1: Progressive Disease | 6 | 9
  Follow-up 2: number analyzed (Participants) | 4 | 5
  Follow-up 2: Complete Response | 3 | 1
  Follow-up 2: Partial Response | 0 | 3
  Follow-up 2: Stable Disease | 0 | 0
  Follow-up 2: Progressive Disease | 1 | 1
  Follow-up 3: number analyzed (Participants) | 1 | 1
  Follow-up 3: Complete Response | 1 | 0
  Follow-up 3: Partial Response | 0 | 0
  Follow-up 3: Stable Disease | 0 | 1
  Follow-up 3: Progressive Disease | 0 | 0
  Follow-up 4: number analyzed (Participants) | 1 | 0
  Follow-up 4: Complete Response | 0 | 0
  Follow-up 4: Partial Response | 1 | 0
  Follow-up 4: Stable Disease | 0 | 0
  Follow-up 4: Progressive Disease | 0 | 0

7. Secondary Outcome: RECIST 1.1 Disease Control Rate by Follow-up Assessment Visit
Description: The proportion of participants with an overall response of Complete Response (CR), Partial Response (PR) and Stable Disease (SD) was reported using investigator assessments per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target, non-target, and new lesions assessed by CT or MRI.
  The timing of follow-up imaging assessments varied depending on how many RLT cycles a participant received. Therefore, regardless of when the imaging assessments occurred, each participant's first follow-up imaging was combined as Follow-up 1, each participant's second follow-up imaging was combined as Follow-up 2, each participant's third follow-up imaging was combined as Follow-up 3, and each participant's fourth follow-up imaging was combined as Follow-up 4.
Time Frame: as for outcome 6
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis
Measure: Number; unit: Percentage of participants
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 28 | 43
Percentage of participants
  Follow-up 1: number analyzed (Participants) | 5 | 12
  Follow-up 1 | 17.9 | 27.9
  Follow-up 2: number analyzed (Participants) | 3 | 4
  Follow-up 2 | 10.7 | 9.3
  Follow-up 3: number analyzed (Participants) | 1 | 1
  Follow-up 3 | 3.6 | 2.3
  Follow-up 4: number analyzed (Participants) | 1 | 0
  Follow-up 4 | 3.6 |

8. Secondary Outcome: Prostate Cancer Working Group 3 (PCWG3) Bone Scan Clinical Impression by Visit
Description: Investigator's assessed bone metastases using the Prostate Cancer Working Group 3 (PCWG3) criteria; new lesions had to be confirmed on a second scan (2+2 rule). The investigator documented their clinical impression of each PCWG3 assessment as Improved, Stable or Progression. The number of participants with a clinical impression of Improved, Stable or Progression according to PCWG3 using investigators assessments was reported by visit.
Time Frame: Screening, Week 8, Week 10, Week 16, Week 18, Week 22, Week 24, Follow-up Week 4, Follow-up Week 6, Follow-up Week 8
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 28 | 43
Participants
  Screening: number analyzed (Participants) | 1 | 0
  Screening: Improved | 0 | 0
  Screening: Stable | 1 | 0
  Screening: Progression | 0 | 0
  Week 8: number analyzed (Participants) | 2 | 6
  Week 8: Improved | 1 | 3
  Week 8: Stable | 1 | 2
  Week 8: Progression | 0 | 1
  Week 10: number analyzed (Participants) | 2 | 4
  Week 10: Improved | 0 | 3
  Week 10: Stable | 2 | 1
  Week 10: Progression | 0 | 0
  Week 16: number analyzed (Participants) | 2 | 2
  Week 16: Improved | 0 | 2
  Week 16: Stable | 2 | 0
  Week 16: Progression | 0 | 0
  Week 18: number analyzed (Participants) | 1 | 3
  Week 18: Improved | 0 | 0
  Week 18: Stable | 0 | 3
  Week 18: Progression | 1 | 0
  Week 22: number analyzed (Participants) | 0 | 1
  Week 22: Improved | 0 | 0
  Week 22: Stable | 0 | 1
  Week 22: Progression | 0 | 0
  Week 24: number analyzed (Participants) | 0 | 1
  Week 24: Improved | 0 | 0
  Week 24: Stable | 0 | 1
  Week 24: Progression | 0 | 0
  Follow-up Week 4: number analyzed (Participants) | 0 | 1
  Follow-up Week 4: Improved | 0 | 0
  Follow-up Week 4: Stable | 0 | 0
  Follow-up Week 4: Progression | 0 | 1
  Follow-up Week 6: number analyzed (Participants) | 0 | 1
  Follow-up Week 6: Improved | 0 | 0
  Follow-up Week 6: Stable | 0 | 0
  Follow-up Week 6: Progression | 0 | 1
  Follow-up Week 8: number analyzed (Participants) | 2 | 0
  Follow-up Week 8: Improved | 0 | 0
  Follow-up Week 8: Stable | 1 | 0
  Follow-up Week 8: Progression | 1 | 0

9. Secondary Outcome: Change From Baseline in Expanded Prostate Cancer Index Composite Short Form (EPIC-26)
Description: The Expanded Prostate Cancer Index-Composite (EPIC) is a well-established patient-reported outcome (PRO) questionnaire developed to monitor health-related quality of life outcomes among prostate cancer. The 26-item version of EPIC, also known as EPIC Short Form or EPIC-26, contains 26 items and 5 domains: Urinary Incontinence (Items 1-4), Urinary Irritative/Obstructive (Items 5-8), Bowel (Items 10-15), Sexual (Items 16-21), and Hormonal (Items 22-26). Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0 to 100 scale for each domain, with higher scores representing better health-related quality of life.
Time Frame: Baseline, Month 3, Month 6, Follow-up Month 3
Population: ITT Population. For each domain, only participants with a value at both baseline and post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 28 | 43
Unit on a scale
  Urinary Incontinence (Baseline): number analyzed (Participants) | 20 | 35
  Urinary Incontinence (Baseline) | 78.3 (26.87) | 77.4 (24.64)
  Urinary Incontinence (Change from BL@Month 3): number analyzed (Participants) | 8 | 9
  Urinary Incontinence (Change from BL@Month 3) | 4.9 (12.57) | 9.7 (20.88)
  Urinary Incontinence (Change from BL@Month 6): number analyzed (Participants) | 3 | 7
  Urinary Incontinence (Change from BL@Month 6) | 11.1 (19.20) | -6.3 (14.66)
  Urinary Incontinence (Change from BL@Follow-up Month 3): number analyzed (Participants) | 0 | 3
  Urinary Incontinence (Change from BL@Follow-up Month 3) |  | -2.1 (9.55)
  Urinary Irritative/Obstructive (Baseline): number analyzed (Participants) | 19 | 35
  Urinary Irritative/Obstructive (Baseline) | 83.2 (20.73) | 84.8 (19.13)
  Urinary Irritative/Obstructive (Change from BL@Month 3): number analyzed (Participants) | 7 | 9
  Urinary Irritative/Obstructive (Change from BL@Month 3) | 17.9 (25.37) | -1.4 (4.17)
  Urinary Irritative/Obstructive (Change from BL@Month 6): number analyzed (Participants) | 3 | 7
  Urinary Irritative/Obstructive (Change from BL@Month 6) | 2.1 (9.55) | 6.3 (8.84)
  Urinary Irritative/Obstructive (Change from BL@Follow-up Month 3): number analyzed (Participants) | 0 | 3
  Urinary Irritative/Obstructive (Change from BL@Follow-up Month 3) |  | 8.3 (9.55)
  Bowel (Baseline): number analyzed (Participants) | 20 | 32
  Bowel (Baseline) | 90.8 (14.60) | 88.4 (14.77)
  Bowel (Change from BL@Month 3): number analyzed (Participants) | 8 | 9
  Bowel (Change from BL@Month 3) | -1.0 (8.55) | 4.0 (18.57)
  Bowel (Change from BL@Month 6): number analyzed (Participants) | 3 | 6
  Bowel (Change from BL@Month 6) | -4.2 (8.33) | 4.9 (16.75)
  Bowel (Change from BL@Follow-up Month 3): number analyzed (Participants) | 0 | 3
  Bowel (Change from BL@Follow-up Month 3) |  | -8.3 (18.16)
  Sexual (Baseline): number analyzed (Participants) | 20 | 33
  Sexual (Baseline) | 8.8 (9.74) | 11.7 (19.66)
  Sexual (Change from BL@Month 3): number analyzed (Participants) | 8 | 9
  Sexual (Change from BL@Month 3) | -4.4 (11.68) | 7.8 (15.76)
  Sexual (Change from BL@Month 6): number analyzed (Participants) | 3 | 7
  Sexual (Change from BL@Month 6) | -4.7 (5.02) | 7.3 (5.82)
  Sexual (Change from BL@Follow-up Month 3): number analyzed (Participants) | 0 | 3
  Sexual (Change from BL@Follow-up Month 3) |  | 4.6 (4.85)
  Hormonal (Baseline): number analyzed (Participants) | 21 | 32
  Hormonal (Baseline) | 77.0 (18.19) | 73.6 (16.13)
  Hormonal (Change from BL@Month 3): number analyzed (Participants) | 8 | 9
  Hormonal (Change from BL@Month 3) | 4.4 (16.35) | 10.4 (24.62)
  Hormonal (Change from BL@Month 6): number analyzed (Participants) | 3 | 7
  Hormonal (Change from BL@Month 6) | 1.7 (28.87) | 10.0 (10.00)
  Hormonal (Change from BL@Follow-up Month 3): number analyzed (Participants) | 0 | 3
  Hormonal (Change from BL@Follow-up Month 3) |  | 8.3 (7.64)

10. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score classifies participants according to their functional impairment, with scores ranging from 0 (fully active) to 5 (dead). ECOG PS: 0 = fully active, able to carry on all pre-disease performance without restriction; 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work; 2 = ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3 = capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5 = dead.
Time Frame: Baseline, Treatment Visit 1, Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Follow-up Month 3, Follow-up Month 12, Follow-up Month 15
Population: ITT Population. Only participants with a value at both baseline and post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
Number analyzed (Participants) | 28 | 43
Scores on a scale
  Baseline: number analyzed (Participants) | 19 | 33
  Baseline | 0.9 (0.81) | 0.9 (0.61)
  Change from BL@Treatment Visit 1: number analyzed (Participants) | 13 | 28
  Change from BL@Treatment Visit 1 | -0.2 (0.60) | 0.0 (0.54)
  Change from BL@Treatment Visit 2: number analyzed (Participants) | 16 | 31
  Change from BL@Treatment Visit 2 | -0.3 (0.60) | -0.1 (0.63)
  Change from BL@Treatment Visit 3: number analyzed (Participants) | 13 | 19
  Change from BL@Treatment Visit 3 | -0.2 (0.73) | -0.2 (0.50)
  Change from BL@Treatment Visit 4: number analyzed (Participants) | 9 | 16
  Change from BL@Treatment Visit 4 | -0.1 (0.93) | -0.3 (0.48)
  Change from BL@Follow-up Month 3: number analyzed (Participants) | 1 | 0
  Change from BL@Follow-up Month 3 | 0.0 (NA) — Only one participant analyzed |
  Change from BL@Follow-up Month 12: number analyzed (Participants) | 0 | 1
  Change from BL@Follow-up Month 12 |  | -1.0 (NA) — Only one participant analyzed
  Change from BL@Follow-up Month 15: number analyzed (Participants) | 0 | 1
  Change from BL@Follow-up Month 15 |  | 0.0 (NA) — Only one participant analyzed

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from informed consent signature through to 24 months after first 177Lu-PSMA-617 treatment therapy.
Description: Any sign or symptom that occurs after written informed consent provided. For TEAE from first dosing (Day 0) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent.
Arm/Group | 177Lu-PSMA-617 (6.0 GBq) | 177Lu-PSMA-617 (7.4 GBq)
All-Cause Mortality (participants affected / at risk) | 3/23 | 3/41
Serious Adverse Events (participants affected / at risk) | 4/23 | 8/41
Other Adverse Events (participants affected / at risk) | 22/23 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 177Lu-PSMA-617 (6.0 GBq) (N=23) | 177Lu-PSMA-617 (7.4 GBq) (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 177Lu-PSMA-617 (6.0 GBq) (N=23) | 177Lu-PSMA-617 (7.4 GBq) (N=41)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 3
Lacrimation increased (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 13
Dry mouth (Gastrointestinal disorders) | 11 | 26
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 18
Saliva altered (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 8
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 13 | 21
Feeling hot (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 3 | 5
Pyrexia (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 2
Parosmia (Nervous system disorders) | 1 | 0
Taste disorder (Nervous system disorders) | 4 | 7
Depression (Psychiatric disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Prostatic pain (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The study began on 05-Jul-17 as an Investigator Initiated Trial and sponsorship was transferred to Endocyte on 01-Jun-18. Recruitment was stopped before the target sample size was achieved based on strategic considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03042312/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03042312/SAP_001.pdf